CLINICAL TRIAL: NCT02166216
Title: The North Sea Race Endurance Exercise Study
Acronym: NEEDED
Status: Active, not recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Nordsjørittet (Unknown); Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: SUS2013ORST01
Record Dates: First submitted 2014-06-11; First posted 2014-06-18 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Prolonged high intensity exercise; Healthy subjects; Cardiovascular risk markers; Troponin; Leisure sports athletes; Cycling; CT coronary angiography; Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum EDTA Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healty subjects: Healthy subjects that participate in a high intensity, endurance bicycle race.

SUMMARY:
Competitions such as marathon running and endurance cycling events are increasingly popular and represent an important motivation for sustaining training among leisure-time athletes. However, there is a concern that prolonged, high-intensity exercise may increase the risk of cardiovascular (CV) events. Following prolonged high-intensity exercise there is an increase in levels of circulating markers of myocardial damage such as Troponin I (TnI). The precise cause and clinical significance of this TnI increase is unknown.

* The primary objective of this study was to determine the relationship between high-sensitive cardiac troponin I (hs-cTnI) levels and coronary artery disease and cardiovascular outcomes in 1000 presumably healthy leisure sport athletes that participated in a 91 km long, high intensity endurance cycling competition.
* The secondary objective was to assess the relationship between other CV risk factors, fitness level and outcomes following high intensity endurance cycling competition in the same population.

DETAILED DESCRIPTION:
The NEEDED observational study was designed to be performed in two phases:

Phase 1 (NEEDED 2013) was a pilot study targeting 100 subjects to test the logistics and identify the optimal blood sampling time points following the race. A total of 97 subjects completed the pilot phase in June 2013.

Phase 2 (NEEDED 2014) aim to recruit another 1000 subjects from the participants of the race in June 2014.

The study populations will be followed for cardiovascular events for up to 20 years following the baseline blood samples.

The results from the two phases will be pooled for the main statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* participants in the "North sea race"
* presumably healthy persons
* signed informed consent
* answered internet based questionnaire prior to the race

Exclusion Criteria:

* cardiac disease
* hypertension
* diabetes mellitus
* use of primary cardiovascular medical prevention

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers participating in the bicycle race "Northsea race" 2013 (pilot) and 2014 (main study), males and females.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-06; Primary Completion 2034-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
The relationship between high sensitive cTni and coronary artery disease and CV events following a high intensity mountain bike competition | 30 days
  Blood will be drawn at 24 hours prior to, and at 3 and 24 hours following a 91 km long mountain bike race. The level of high sensitive TnI will be analyzed at all time-points. All study participants will be followed-up for 30 days, and all events will be recorded. Additionally, based on data from the NEEDED 2013 pilot study all participants with an increase in high sensitive cTni > 200 ng/l within 24 hours following the cycling competition will be assessed by CT coronary angiography within the first week following the race to determine the presence of significant coronary artery disease in order to detect subclinical coronary artery disease.

SECONDARY OUTCOMES:
The relationship between high sensitive cTni and coronary artery disease and CV events following a high intensity mountain bike competition | 1 year
  Blood will be drawn at 24 hours prior to, and at 3 and 24 hours following a 91 km long mountain bike race. The level of high sensitive TnI will be analyzed at all timepoints.All study participants will be followed-up for 30 days, and all CV events will be recorded. Additionally, based on data from the NEEDED 2013 pilot study all participants with an increase in high sensitive cTni > 200 ng/l within 24 hours following the cycling competition will be assessed by CT coronary angiography within the first week following the race to determine the presence of significant coronary artery disease in order to detect subclinical coronary artery disease.
The relationship between high sensitive cTni and coronary artery disease and CV events following a high intensity mountain bike competition | 5 years
  Blood will be drawn at 24 hours prior to, and at 3 and 24 hours following a 91 km long mountain bike race. The level of high sensitive TnI will be analyzed at all timepoints.All study participants will be followed-up for 30 days, and all CV events will be recorded. Additionally, based on data from the NEEDED 2013 pilot study all participants with an increase in high sensitive cTni > 200 ng/l within 24 hours following the cycling competition will be assessed by CT coronary angiography within the first week following the race to determine the presence of significant coronary artery disease in order to detect subclinical coronary artery disease.
The relationship between high sensitive cTni and coronary artery disease and CV events following a high intensity mountain bike competition | 20 years
  Blood will be drawn at 24 hours prior to, and at 3 and 24 hours following a 91 km long mountain bike race. The level of high sensitive TnI will be analyzed at all time-points. All study participants will be followed-up for 30 days, and all CV events will be recorded. Additionally, based on data from the NEEDED 2013 pilot study all participants with an increase in high sensitive cTni > 200 ng/l within 24 hours following the cycling competition will be assessed by CT coronary angiography within the first week following the race to determine the presence of significant coronary artery disease in order to detect subclinical coronary artery disease.

CONTACTS AND LOCATIONS:
Overall Officials: Stein Ørn, MD PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Derived] Erevik CB, Kleiven O, Froysa V, Bjorkavoll-Bergseth M, Chivulescu M, Klaeboe LG, Dejgaard L, Auestad B, Skadberg O, Melberg T, Urheim S, Haugaa K, Edvardsen T, Orn S. Exercise-Induced Cardiac Troponin I Elevation Is Associated With Regional Alterations in Left Ventricular Strain in High-Troponin Responders. J Am Heart Assoc. 2024 Aug 20;13(16):e034382. doi: 10.1161/JAHA.124.034382. Epub 2024 Aug 19. PMID 39158569
- [Derived] Bjorkavoll-Bergseth M, Erevik CB, Kleiven O, Eijsvogels TMH, Skadberg O, Froysa V, Wiktorski T, Auestad B, Edvardsen T, Aakre KM, Orn S. Determinants of Interindividual Variation in Exercise-Induced Cardiac Troponin I Levels. J Am Heart Assoc. 2021 Sep 7;10(17):e021710. doi: 10.1161/JAHA.121.021710. Epub 2021 Aug 28. PMID 34459237
- [Derived] Hansen MW, Orn S, Erevik CB, Bjorkavoll-Bergseth MF, Skadberg O, Melberg TH, Aakre KM, Kleiven O. Regular consumption of cod liver oil is associated with reduced basal and exercise-induced C-reactive protein levels; a prospective observational trial : A NEEDED (The North Sea Race Endurance Exercise Study) 2014 sub-study. J Int Soc Sports Nutr. 2021 Jun 28;18(1):51. doi: 10.1186/s12970-021-00437-1. PMID 34183020
- [Derived] Skranes JB, Kleiven O, Aakre KM, Skadberg O, Melberg TH, Omland T, Orn S. High-Sensitivity Cardiac Troponin I and T Response Following Strenuous Activity is Attenuated by Smokeless Tobacco: NEEDED (North Sea Race Endurance Exercise Study) 2014. J Am Heart Assoc. 2020 Oct 20;9(19):e017363. doi: 10.1161/JAHA.120.017363. Epub 2020 Sep 15. PMID 32930023
- [Derived] Bjorkavoll-Bergseth M, Kleiven O, Auestad B, Eftestol T, Oskal K, Nygard M, Skadberg O, Aakre KM, Melberg T, Gjesdal K, Orn S. Duration of Elevated Heart Rate Is an Important Predictor of Exercise-Induced Troponin Elevation. J Am Heart Assoc. 2020 Feb 18;9(4):e014408. doi: 10.1161/JAHA.119.014408. Epub 2020 Feb 17. PMID 32065043
- [Derived] Kleiven O, Omland T, Skadberg O, Melberg TH, Bjorkavoll-Bergseth MF, Auestad B, Bergseth R, Greve OJ, Aakre KM, Orn S. Race duration and blood pressure are major predictors of exercise-induced cardiac troponin elevation. Int J Cardiol. 2019 May 15;283:1-8. doi: 10.1016/j.ijcard.2019.02.044. Epub 2019 Feb 23. PMID 30842026